CLINICAL TRIAL: NCT06828939
Title: Pulmonary Vein Isolation With the Single Shot Endoscopic Ultra-Compliant Pulsed Field Ablation Balloon for the Treatment of Atrial Fibrillation
Brief Title: Pulmonary Vein Isolation With the Single Shot Endoscopic Ultra-Compliant PFA Balloon for the Treatment of AF
Acronym: VISION AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CardioFocus (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-6073
Record Dates: First submitted 2025-02-04; First posted 2025-02-17 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Atrial Fibrillation (Paroxysmal)
Keywords: ablation; pulsed field ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: OptiShot PFA Balloon System
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Treatment Arm (Experimental): The treatment arm will undergo catheter ablation for symptomatic paroxysmal atrial fibrillation with the OptiShot Pulsed Field Ablation (PFA) Balloon System
  Interventions: Device: pulsed field ablation

INTERVENTIONS:
Device: pulsed field ablation — Pulsed field ablation using a ultra-compliant endoscopic PFA balloon.

SUMMARY:
This is a prospective, single-arm First-in-Human study to demonstrate the safety and effectiveness of the CardioFocus OptiShot Pulsed Field Ablation System for catheter ablation of atrial fibrillation (AF). Patients with symptomatic paroxysmal (short-duration) AF who have not had a previous catheter ablation for AF will be considered for the study. Patients will be followed for one year after the initial ablation procedure.

DETAILED DESCRIPTION:
This is a prospective, single-arm First-in-Human study to demonstrate the safety and effectiveness of the CardioFocus OptiShot Pulsed Field Ablation System for catheter ablation of atrial fibrillation (AF). Patients with symptomatic paroxysmal AF who are undergoing first-time pulmonary vein isolation will be considered for the study. Patients will be followed for one year after the initial ablation procedure.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent symptomatic PAF with at least one documented episode
* Failure or intolerance of at least one AAD
* Age 18-75 years
* Patient is indicated for an ablation procedure according to society guidelines or study site practice
* Patient is willing and able to give informed consent/participate in baseline and follow-up assessments for the duration of the study

Exclusion Criteria:

* overall good health as established by multiple criteria

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint - Acute Procedure Success | During procedure
  Pulmonary vein isolation at the end of the index procedure
Primary Safety Endpoint - Rate of Primary Serious Adverse Events | 7 days (unless otherwise specified)
  The rate of participants with at least 1 of the following Primary Serious Adverse Events occurring within 7 days unless otherwise specified:
  * AE fistula (assessed at >=60 days)
  * Cardiac perforation, tamponade, or pericardial effusion
  * Complete heart block
  * Death
  * Major vascular access complications/bleeding requiring surgical intervention or blood transfusion
  * MI
  * Pericarditis
  * PNI resulting in persistent diaphragmatic paralysis (assessed at <=60 days)
  * PV stenosis (assessed at <=60 days)
  * Stroke/CVA
  * Thromboembolism
  * TIA
  * Vagal nerve injury/gastroparesis

SECONDARY OUTCOMES:
Secondary Effectiveness Endpoint - Chronic Durability | 90 days
  Percentage of treated PVs with documented PVI at the remapping procedure
Secondary Effectiveness Endpoint - 12-Month Freedom from Atrial Arrhythmia | 12 months
  Freedom from documented atrial arrhythmia (AF/AFL/AT) episodes of > 30 seconds duration after 60-day blanking period documented by TTM or Holter monitor

CONTACTS AND LOCATIONS:
Locations (1):
- Na Homolce Hospital, Prague, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: No